CLINICAL TRIAL: NCT03069690
Title: Optimizing Health From Pregnancy Through One Year Postpartum: A Sequential Multiple Assignment Randomized Trial (SMART) of Perinatal Lifestyle Interventions
Brief Title: Optimizing Health From Pregnancy Through One Year Postpartum
Acronym: HABIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Michele Levine, Professor, University of Pittsburgh
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PRO16020497; R01HL132578-01 (NIH)
Record Dates: First submitted 2017-02-20; First posted 2017-03-03 (Actual); Results first posted 2025-04-16 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-03

CONDITIONS: Obesity; Pregnancy Related
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: The intervention model is a nonrestricted sequential multiple assignment randomized trial (SMART). Participants are randomized to intervention or control during pregnant and again postpartum.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- HABITpreg; TAUpost (Experimental): Participants will receive study intervention during pregnant and treatment as usual postpartum.
  Interventions: Behavioral: HABITpreg
- HABITpreg, HABITpost (Experimental): Participants will receive study intervention during pregnancy and study intervention during the postpartum period.
  Interventions: Behavioral: HABITpreg; Behavioral: HABITpost
- TAUpreg; HABITpost (Experimental): Participants will receive treatment as usual during pregnancy and study intervention during the postpartum period.
  Interventions: Behavioral: HABITpost
- TAUpreg; TAUpost (No Intervention): Participates will receive treatment as usual during pregnancy and treatment as usual during the postpartum period.

INTERVENTIONS:
Behavioral: HABITpreg — Treatment during pregnancy will consist of up to 10 in person sessions taking place at regularly scheduled obstetric appointments, at the investigator's research building, or a nearby location. Participants in the HABITpregnancy group will also receive texts and phone calls between sessions. HABIT will focus on weight, physical activity, eating and psychosocial issues. Women will receive consultation about nutritional balance, dietary guidelines for pregnant women and advice to maintain an optimal rate of weight gain according to prepregnancy BMI. Women will use self-monitoring forms to identify and modify cues for unhealthy behaviors. Beliefs about body weight and eating during pregnancy will be addressed and effects of physical activity on body weight, health, and mood will be included.
  Due to COVID-19(coronavirus disease) restrictions and safety guidelines, HABIT pregnant treatment sessions have been taking place virtually, using video chat or phone calls starting in March 2020.
  Arms: HABITpreg, HABITpost; HABITpreg; TAUpost
Behavioral: HABITpost — Treatment during the postpartum period (HABITpost) will consist of an intervention over the 24 weeks immediately following delivery. Treatment will include 12 biweekly sessions completed over the phone or in person. In person sessions will be done at the participant's home or another convenient location. Additionally, participants will receive calls and texts between sessions. Sessions will focus on weight, physical activity, eating and psychosocial issues.
  Due to COVID-19 restrictions and safety guidelines, HABIT post treatment sessions have been taking place virtually, using video chat or phone calls starting in March 2020.
  Arms: HABITpreg, HABITpost; TAUpreg; HABITpost

SUMMARY:
This study will evaluate the impact of different combinations of intervention as a function of gestational weight gain in pregnant woman. Participants will be randomized at two points during the study. Participants will first be randomized at enrollment to receive study intervention during pregnancy or treatment as usual. Participants will also be randomized just before delivery to receive intervention postpartum or treatment as usual.

DETAILED DESCRIPTION:
The perinatal period, from pregnancy through the first postpartum year, has important implications for women's health. Excessive gestational weight gain is linked to deleterious health outcomes; yet most women exceed guidelines established for gestational weight gain , particularly women who begin pregnancy overweight or obese. These women are likely to remain overweight or obese at one year postpartum even if gestational weight gain is within guidelines and pregnancy-related weight gain is lost postpartum. Efforts to mitigate the health risks related to perinatal overweight can have substantial benefits for women's longer-term obesity and cardiometabolic health. To date, interventions to minimize excessive gestational weight gain alone have had limited impact. Some women may require continued intervention in the postpartum period to achieve optimal weight management. Alternatively, intervention delivered only postpartum may be sufficient to achieve a healthier weight at one year postpartum. It also is important to adapt intervention as women's needs vary over the course of pregnancy and postpartum. Accordingly, this application proposes a sequential multiple assignment randomized trial (SMART) to determine the efficacy of different intervention sequences during pregnancy, postpartum, or both. This non-restricted SMART also will allow investigators to investigate the impact of different combinations of intervention as a function of gestational weight gain. The proposed SMART is innovative as the first effort to evaluate different sequences of intervention across the perinatal period to mitigate maternal health risk by one year postpartum.

Pregnant women (N=300), stratified by prenatal weight status (body mass index=25-29.9 vs. ≥30) will be enrolled at entry into prenatal care and randomized initially to intervention that addresses the challenges of weight and self-regulation during pregnancy, Health and Behaviors in Transition (HABITpreg), or an educationally-enhanced treatment as usual (TAUpreg). At delivery, women will be re-randomized to a postpartum self-regulation intervention (HABITpost) or educationally-enhanced treatment as usual (TAUpost). Women will complete assessments at a prenatal baseline, the end of pregnancy, and 6- and 12-months postpartum.

ELIGIBILITY:
Inclusion Criteria:

* Have a prenatal BMI ≥ 25
* Are at or before 18 weeks and 4 days of gestation
* Are English speaking
* Have a singleton pregnancy

Exclusion Criteria:

* Multiple gestations
* Preexisting diabetes
* Previous bariatric surgery in the previous 3 years
* Use of medications known to affect weight (e.g., second generation antipsychotic medications, regular steroid use).
* Women who endorse acute psychiatric symptoms (e.g., suicidality) that warrant immediate treatment will be excluded and referred for care.

Min Age: 14 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2024-01-25 (Actual); Study Completion 2024-06-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michele Levine, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment for the project began in January, 2017 and the first participant was enrolled on February 1, 2017. Enrollment of pregnant individuals into this clinical trial concluded in September 2022.
Pre-assignment Details: Prior to pregnancy randomization:
  3 participants had pregnancy loss. 5 participants never completed their baseline assessment and were not eligible to be randomized.
Groups:
- TAUpreg: Participants will receive treatment as usual during pregnancy
- HABITpreg; TAUpost: Participants will receive study intervention during pregnant and treatment as usual postpartum.
  HABITpreg: Treatment during pregnancy will consist of up to 10 in person sessions taking place at regularly scheduled obstetric appointments, at the investigator's research building, or a nearby location. Participants in the HABITpregnancy group will also receive texts and phone calls between sessions. HABIT will focus on weight, physical activity, eating and psychosocial issues. Women will receive consultation about nutritional balance, dietary guidelines for pregnant women and advice to maintain an optimal rate of weight gain according to prepregnancy BMI. Women will use self-monitoring forms to identify and modify cues for unhealthy behaviors. Beliefs about body weight and eating during pregnancy will be addressed and effects of physical activity on body weight, health, and mood will be included.
  Due to COVID-19(coronavirus disease) restrictions and safety guidelines, HABIT pregnant treatment sessions have been taking place virtually, using video chat or phone calls starting in March 2020.
- HABITpreg, HABITpost: Participants will receive study intervention during pregnancy and the postpartum period.
  HABITpreg: Treatment during pregnancy will consist of up to 10 in person sessions taking place at regularly scheduled obstetric appointments, at the investigator's research building, or a nearby location. Participants will also receive texts and phone calls between sessions. HABIT will focus on weight, physical activity, eating and psychosocial issues. Women will receive consultation about nutritional balance, dietary guidelines for pregnant women and advice to maintain an optimal rate of weight gain according to prepregnancy BMI. Women will use self-monitoring forms to identify and modify cues for unhealthy behaviors. Beliefs about body weight and eating during pregnancy will be addressed and effects of physical activity on body weight, health, and mood will be included.
  HABITpost: Treatment during the postpartum period will consist of an intervention over the 24 weeks immediately following delivery. Treatment will include 12 biweekly sessions completed over the phone or in person. In person sessions will be done at the participant's home or another convenient location. Participants will receive calls and texts between sessions. Sessions will focus on weight, physical activity, eating and psychosocial issues.
  Due to COVID-19 restrictions and safety guidelines, treatment sessions have been taking place virtually, using video chat or phone calls starting in March 2020.
- TAUpreg; HABITpost: Participants will receive treatment as usual during pregnancy and study intervention during the postpartum period.
  HABITpost: Treatment during the postpartum period (HABITpost) will consist of an intervention over the 24 weeks immediately following delivery. Treatment will include 12 biweekly sessions completed over the phone or in person. In person sessions will be done at the participant's home or another convenient location. Additionally, participants will receive calls and texts between sessions. Sessions will focus on weight, physical activity, eating and psychosocial issues.
  Due to COVID-19 restrictions and safety guidelines, HABIT post treatment sessions have been taking place virtually, using video chat or phone calls starting in March 2020.
Period: Pregnancy Intervention
Arm/Group | HABITpreg | TAUpreg | HABITpreg; TAUpost | HABITpreg, HABITpost | TAUpreg; HABITpost | TAUpreg; TAUpost
Started | 25 | 18 | 64 | 67 | 70 | 68
Completed | 0 | 0 | 64 | 67 | 70 | 68
Not Completed | 25 | 18 | 0 | 0 | 0 | 0
Not completed — Pregnancy loss | 9 | 4 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 16 | 14 | 0 | 0 | 0 | 0
Period: Postpartum Intervention
Arm/Group | HABITpreg | TAUpreg | HABITpreg; TAUpost | HABITpreg, HABITpost | TAUpreg; HABITpost | TAUpreg; TAUpost
Started | 0 | 0 | 64 | 67 | 70 | 68
Completed | 0 | 0 | 59 | 62 | 68 | 64
Not Completed | 0 | 0 | 5 | 5 | 2 | 4
Not completed — Lost to Follow-up | 0 | 0 | 5 | 5 | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HABITpreg | TAUpreg | HABITpreg; TAUpost | HABITpreg, HABITpost | TAUpreg; HABITpost | TAUpreg; TAUpost | Total
Number analyzed (Participants) | 25 | 18 | 64 | 67 | 70 | 68 | 312
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.55 (6.21) | 28.86 (4.16) | 31.01 (5.09) | 30.83 (4.17) | 31.31 (4.86) | 31.26 (5.13) | 31.11 (4.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 18 | 64 | 67 | 70 | 68 | 312
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 2 | 4 | 3 | 2 | 15
  Not Hispanic or Latino | 24 | 15 | 62 | 63 | 66 | 66 | 296
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 2 | 0 | 1 | 0 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Black or African American | 9 | 9 | 11 | 17 | 14 | 17 | 77
  White | 13 | 5 | 48 | 47 | 55 | 46 | 214
  More than one race | 2 | 3 | 3 | 2 | 0 | 5 | 15
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Maternal Weight
Description: Maternal weight in lbs
Time Frame: Baseline and 1 year postpartum
Population: Missing T12 weight data from 17 participants. (HABITpreg; TAUpost- missing 5, HABITpreg; HABITpost- missing 5, TAUpreg; HABITpost- missing 2, TAUpreg; TAUpost- missing 5)
  As discussed in the flow, participants in the HABITpreg (25) and TAUpreg (18) did not complete the second randomization therefore we only have baseline data for these individuals.
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | HABITpreg | TAUpreg | HABITpreg; TAUpost | HABITpreg, HABITpost | TAUpreg; HABITpost | TAUpreg; TAUpost
Number analyzed (Participants) | 25 | 18 | 64 | 67 | 70 | 68
pounds
  12 month follow-up: number analyzed (Participants) | 0 | 0 | 59 | 62 | 68 | 63
  12 month follow-up |  |  | 196.59 (44.81) | 201.03 (43.64) | 193.70 (37.51) | 201.66 (45.54)
  Baseline | 202.16 (42.10) | 217.09 (54.92) | 194.16 (40.33) | 196.73 (39.44) | 190.13 (32.84) | 195.62 (41.32)
Statistical Analysis 1: Comparison: TAUpreg; HABITpost; Test type: Superiority; p = .80, ANCOVA — The value was not adjusted for multiple comparisons; Mean Difference (Net) = -0.3996, 95% CI 2-sided [-5.649 to 4.850], Standard Error of Mean 2.665
Statistical Analysis 2: Comparison: HABITpreg; TAUpost; Test type: Superiority; p = .80, ANCOVA — The value was not adjusted for multiple comparisons; Mean Difference (Net) = -3.3870, 95% CI 2-sided [-8.813 to 2.039], Standard Error of Mean 2.755
Statistical Analysis 3: Comparison: HABITpreg, HABITpost; Test type: Superiority; p = .80, ANCOVA — The value was not adjusted for multiple comparisons; Mean Difference (Net) = -1.1729, 95% CI 2-sided [-6.530 to 4.184], Standard Error of Mean 2.720

2. Secondary Outcome: Maternal Lipids
Description: Blood Analysis of Maternal Lipids (High-Density Lipoprotein (HDL), Low-Density Lipoprotein calculated (LDL), Cholesterol, Triglyceride).
Time Frame: Baseline and 1 year postpartum (T12)
Population: Missing blood samples from 36 participants at T12 follow-up (HABITpreg; TAUpost- missing 9, HABITpreg; HABITpost- missing 11; TAUpreg; HABITpost- missing 7, TAUpreg; TAUpost- missing 9)
  Missing 1 sample at baseline in the TAUpreg; TAUpost group.
  As discussed in the flow, participants in the HABITpreg (25) and TAUpreg (18) did not complete the second randomization therefore we only have baseline data for these individuals.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | HABITpreg | TAUpreg | HABITpreg; TAUpost | HABITpreg, HABITpost | TAUpreg; HABITpost | TAUpreg; TAUpost
Number analyzed (Participants) | 25 | 18 | 64 | 67 | 70 | 68
mg/dL
  High-Density Lipoprotein- T12 follow-up: number analyzed (Participants) | 0 | 0 | 55 | 56 | 63 | 59
  High-Density Lipoprotein- T12 follow-up |  |  | 55.16 (11.69) | 53.77 (13.64) | 55.57 (10.92) | 54.29 (11.38)
  Low-Density Lipoprotein calculated- T12 follow-up: number analyzed (Participants) | 0 | 0 | 55 | 56 | 63 | 59
  Low-Density Lipoprotein calculated- T12 follow-up |  |  | 97.67 (27.15) | 103.63 (32.52) | 106.10 (33.40) | 104.00 (33.80)
  Cholesterol- T12 follow-up: number analyzed (Participants) | 0 | 0 | 55 | 56 | 63 | 59
  Cholesterol- T12 follow-up |  |  | 175.62 (35.95) | 178.75 (42.79) | 180.59 (32.84) | 177.75 (41.31)
  Triglyceride- T12 follow-up: number analyzed (Participants) | 0 | 0 | 55 | 56 | 63 | 59
  Triglyceride- T12 follow-up |  |  | 113.87 (71.66) | 106.79 (69.02) | 94.51 (48.36) | 96.97 (49.11)
  High-Density Lipoprotein- Baseline: number analyzed (Participants) | 25 | 18 | 64 | 67 | 70 | 67
  High-Density Lipoprotein- Baseline | 66.84 (12.25) | 60.28 (15.11) | 64.94 (11.44) | 62.21 (13.43) | 65.53 (12.93) | 66.27 (11.70)
  Low-Density Lipoprotein calculated- Baseline: number analyzed (Participants) | 25 | 18 | 64 | 67 | 70 | 67
  Low-Density Lipoprotein calculated- Baseline | 99.16 (22.50) | 84.50 (21.89) | 96.77 (26.16) | 100.61 (33.46) | 102.57 (27.99) | 99.99 (27.20)
  Cholesterol- Baseline: number analyzed (Participants) | 25 | 18 | 64 | 67 | 70 | 67
  Cholesterol- Baseline | 188.08 (27.75) | 165.33 (28.75) | 187.47 (32.96) | 187.52 (43.20) | 191.74 (36.14) | 189.33 (34.65)
  Triglyceride- Baseline: number analyzed (Participants) | 25 | 18 | 64 | 67 | 70 | 67
  Triglyceride- Baseline | 110.80 (39.54) | 102.78 (43.60) | 128.79 (54.53) | 123.24 (54.70) | 118.06 (54.37) | 115.72 (41.55)

3. Secondary Outcome: Maternal Inflammatory Markers
Description: Maternal inflammatory markers from blood analysis
Time Frame: Baseline and 1 year postpartum (T12)
Population: Blood analysis for maternal inflammatory markers have not been completed, and will not be run in the future, due to prohibitive costs associated with the assays.
Arm/Group | HABITpreg; TAUpost | HABITpreg, HABITpost | TAUpreg; HABITpost | TAUpreg; TAUpost
Number analyzed (Participants) | 0 | 0 | 0 | 0

4. Secondary Outcome: Depressive Symptoms (EPDS)
Description: Scores from the Edinburgh Postnatal Depression Scale (EPDS)
  This scale is developed to assist health professionals in detecting mothers suffering from postpartum depression (PPD), consists of 10 short statements indicating how a mother felt during the previous week. Each response is scored 0, 1, 2 and 3 based on the seriousness of the symptom. The total score is found by adding together the scores for each of the 10 items. Scores range from 0-30. Scoring above 12 or 13 are likely to be suffering from depression and should seek medical attention. A careful clinical evaluation by a health care professional is needed to confirm a diagnosis and establish a treatment plan.
Time Frame: Baseline and 1 year postpartum (T12)
Population: At T12 follow-up- Scores from 24 participants are missing due to incomplete data on them at T12. (HABITpreg; TAUpost- 7 missing, HABITpreg; HABITpost- 6 missing, TAUpreg; HABITpost- 4 missing, TAUpreg; TAUpost- 7 missing)
  As discussed in the flow, participants in the HABITpreg (25) and TAUpreg (18) did not complete the second randomization therefore we only have baseline data for these individuals.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HABITpreg | TAUpreg | HABITpreg; TAUpost | HABITpreg, HABITpost | TAUpreg; HABITpost | TAUpreg; TAUpost
Number analyzed (Participants) | 25 | 18 | 64 | 67 | 70 | 68
score on a scale
  T12 follow-up: number analyzed (Participants) | 0 | 0 | 57 | 61 | 66 | 61
  T12 follow-up |  |  | 5.28 (5) | 4.70 (5.23) | 5.83 (6.19) | 7.03 (6.79)
  Baseline | 6.08 (5.56) | 8.61 (6.12) | 6.13 (4.77) | 4.93 (4.68) | 5.61 (5.33) | 6.47 (4.89)

5. Secondary Outcome: Depressive Symptoms (CESD)
Description: Scores from the Center for Epidemiological Studies-Depression (CESD)
  This scale is a self-report measure of depression. Questions measure 8 different subscales, including: Sadness (Dysphoria): (Q. 2, 4, 6), Loss of Interest (Anhedonia): (Q. 8, 10), Appetite: (Q. 1, 18), Sleep: (Q. 5, 11, 19), Thinking / concentration: (Q. 3, 20), Guilt (Worthlessness): (Q. 9, 17), Tired (Fatigue): (Q. 7, 16), Movement (Agitation): (Q. 12, 13), Suicidal Ideation: (Q. 14, 15) Each response is scored 0, 1, 2 and 3 based on the frequency of the symptom. The total score is calculated by finding the sum of 20 items. Scores range from 0-60. A score equal to or above 16 indicates a person at risk for clinical depression.
Time Frame: Baseline and 1 year postpartum (T12)
Population: At T12 follow-up- Scores from 21 participants are missing due to incomplete data on them at T12. (HABITpreg; TAUpost- 7 missing, HABITpreg; HABITpost- 5 missing, TAUpreg; HABITpost- 5 missing, TAUpreg; TAUpost- 4 missing)
  As discussed in the flow, participants in the HABITpreg (25) and TAUpreg (18) did not complete the second randomization therefore we only have baseline data for these individuals.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HABITpreg | TAUpreg | HABITpreg; TAUpost | HABITpreg, HABITpost | TAUpreg; HABITpost | TAUpreg; TAUpost
Number analyzed (Participants) | 25 | 18 | 64 | 67 | 70 | 68
score on a scale
  T12 follow-up: number analyzed (Participants) | 0 | 0 | 57 | 62 | 65 | 64
  T12 follow-up |  |  | 11.68 (10.70) | 10.29 (9.52) | 12.78 (11.70) | 13.25 (11.49)
  Baseline | 13.88 (10.63) | 18.22 (11.24) | 13.19 (9.14) | 11.06 (8.31) | 12.04 (8.90) | 13.18 (8.61)

6. Other Pre Specified Outcome: Gestational Weight Gain
Description: Gestational weight gain in lbs
Time Frame: Time of delivery
Population: Missing weight data from 17 participants. (HABITpreg; TAUpost- missing 5, HABITpreg; HABITpost- missing 5, TAUpreg; HABITpost- missing 2, TAUpreg; TAUpost- missing 5)
  As discussed in the flow, participants in the HABITpreg (25) and TAUpreg (18) did not complete the second randomization therefore we only have baseline data for these individuals.
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | HABITpreg | TAUpreg | HABITpreg; TAUpost | HABITpreg, HABITpost | TAUpreg; HABITpost | TAUpreg; TAUpost
Number analyzed (Participants) | 0 | 0 | 59 | 62 | 68 | 63
pounds |  |  | 6.32 (19.41) | 7.14 (16.02) | 7.63 (16.52) | 10.76 (16.91)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over the course of the study. Throughout pregnancy and through 1 year postpartum.
Groups:
- HABITpreg: Participants will receive study intervention during pregnancy.
- HABITpreg; TAUpost: Participants will receive study intervention during pregnancy and treatment as usual postpartum.
  HABITpreg: Treatment during pregnancy will consist of up to 10 in person sessions taking place at regularly scheduled obstetric appointments, at the investigator's research building, or a nearby location. Participants in the HABITpregnancy group will also receive texts and phone calls between sessions. HABIT will focus on weight, physical activity, eating and psychosocial issues. Women will receive consultation about nutritional balance, dietary guidelines for pregnant women and advice to maintain an optimal rate of weight gain according to prepregnancy BMI. Women will use self-monitoring forms to identify and modify cues for unhealthy behaviors. Beliefs about body weight and eating during pregnancy will be addressed and effects of physical activity on body weight, health, and mood will be included.
  Due to COVID-19(coronavirus disease) restrictions and safety guidelines, HABIT pregnant treatment sessions have been taking place virtually, using video chat or phone calls starting in March 2020.
Arm/Group | HABITpreg | TAUpreg | HABITpreg; TAUpost | HABITpreg, HABITpost | TAUpreg; HABITpost | TAUpreg; TAUpost
All-Cause Mortality (participants affected / at risk) | 0/156 | 0/156 | 0/64 | 0/67 | 0/70 | 0/68
Serious Adverse Events (participants affected / at risk) | 0/156 | 0/156 | 0/64 | 0/67 | 0/70 | 0/68
Other Adverse Events (participants affected / at risk) | 9/156 | 4/156 | 0/64 | 0/67 | 0/70 | 0/68
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HABITpreg (N=156) | TAUpreg (N=156) | HABITpreg; TAUpost (N=64) | HABITpreg, HABITpost (N=67) | TAUpreg; HABITpost (N=70) | TAUpreg; TAUpost (N=68)
Pregnancy loss (Pregnancy, puerperium and perinatal conditions) | 9 (9) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-11-20): https://cdn.clinicaltrials.gov/large-docs/90/NCT03069690/Prot_SAP_000.pdf